CLINICAL TRIAL: NCT04917705
Title: Search for Diagnostic and Prognostic Biomarkers (Molecular Signatures) in Systemic Sclerosis and Inflammatory Myopathies by a Multi-OMIC Strategy Integrating a Single Cell Analysis Approach
Brief Title: Search for Diagnostic and Prognostic Biomarkers in Systemic Sclerosis and Inflammatory Myopathies
Acronym: SCLEROMYOMICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8181
Record Dates: First submitted 2021-04-22; First posted 2021-06-08 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Systemic Sclerosis; Inflammatory Myopathies
Keywords: Scleroderma; Myopathy; Multi-OMICS; Biomarkers; Single-cell
MeSH Terms: conditions — Scleroderma, Systemic; Myositis; Scleroderma, Diffuse; Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of biological samples — Skin, muscle fiber and blood sampling

SUMMARY:
Systemic sclerosis and inflammatory myopathies, which sometimes combine (scleromyositis), have shared pathophysiological elements. In both diseases, many cell subtypes are involved in damage to organs such as T lymphocytes, B lymphocytes, and unconventional (non-B, non-T) lymphocytes called innate lymphoid cell (ILC). The increasing complexity of our understanding of the immune system (multiplication of recognized cell subtypes) also makes the strategies for analyzing pathophysiological mechanisms more complex. Currently, no biomarker perfectly predicts the phenotype and evolution of patients. Multi-OMIC analyzes will be performed (identification of cell populations as well as genomic, transcriptomic and proteomic characterization) in blood and tissue samples (skin and muscle biopsy) in patients with systemic sclerosis and inflammatory myopathies, with the objective of identifying discriminating molecular signatures (biomarkers) according to the characteristics of the disease and its evolution.

DETAILED DESCRIPTION:
Cohort study, monocentric, comparative, non-randomized, open-label, prospective and longitudinal, quasi-experimental.

Participating subjects will be classified according to their clinical, biological and additional investigations into one of the 4 populations presented in the eligibility criteria.

A 1st sampling point will be carried out at inclusion visit (baseline). Prospective follow-up of participating patients will be carried out as part of their routine care (1 to 2 visits per year or more if disease complications appear).

During the 5-year follow-up, the investigating physician will remain attentive to the appearance of a new clinical element which will mark the course of the disease.

During the follow-up, 2 more sampling points will be carried out (blood and / or skin) on each participating patient.

Blood samples and muscle biopsies will be carried out in the usual way during diagnostic and therapeutic management. An additional volume of blood, an additional muscle biopsy (on the occasion of the one performed for diagnosis) and two superficial skin biopsies (1 sclerotic tissue & 1 healthy tissue) will be taken for research purposes.

Inclusion in this cohort will not change the management of the patient, either with regard to his treatment or his follow-up.

Multi-omics analyzes will include single cell RNAseq, as well as proteomics and genomics analysis:

* Transcriptomic analysis will be performed on PMBC, muscle and skin.
* Genomic analysis (exome & whole genome) will be performed on PMBC, muscle and skin.
* Proteomic analysis will be performed on serum, PMBC, muscle and skin.
* Single cell analysis will be performed on PMBC, muscle and skin. During the analysis, the clinical characteristics of baseline, the treatments and the evolutions during the follow-up will be compared to reveal the clinical relevance of the multi-OMIC signatures.

ELIGIBILITY:
Inclusion Criteria:

* Control population without inflammatory myopathy (population 1), suspected myopathy for whom a blood test and muscle biopsy are required to confirm the diagnosis
* Confirmed inflammatory myopathy (population 2)
* Control population without systemic sclerosis (population 3), with primary Raynaud's phenomenon
* Early diffuse systemic cutaneous scleroderma (population 4)
* Male or female (age ≥ 18, no upper age limit)

Exclusion Criteria:

Populations 1 & 2

* Contraindication to muscle biopsy
* Diagnosed for another neuromuscular disease
* Taking an immunosuppressant / immunomodulator treatment within 3 months before inclusion
* Unbalanced cardiovascular pathology

Population 3 & 4

* Contraindication to skin biopsy
* Capillaroscopic and / or immunological anomaly suggesting scleroderma
* Suspicion of scleroderma but diagnosed for another connectivitis
* Immunosuppressive treatment (corticosteroids> 15 mg, methotrexate, mycophenolate mofetil) introduced for more than 1 month
* Active or recent cancer <3 years (apart from non-melanoma skin cancer).

For all

- Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Evolution of the molecular profiles (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing]) of systemic sclerosis during 5 years. | At Day 1
  This study is descriptive (non-analytical), without prior hypothesis. Molecular profiles will be assessed by integration of multi-OMIC tools from a wide range of areas of biochemistry, chemistry, physics, computing science and molecular biology.
  During the 5-year follow-up, the investigating physician will remain attentive to the appearance of a new clinical element which will mark the course of the systemic sclerosis.
Evolution of the molecular profiles (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing]) of systemic sclerosis during 5 years. | At 12 months
  This study is descriptive (non-analytical), without prior hypothesis. Molecular profiles will be assessed by integration of multi-OMIC tools from a wide range of areas of biochemistry, chemistry, physics, computing science and molecular biology.
  During the 5-year follow-up, the investigating physician will remain attentive to the appearance of a new clinical element which will mark the course of the systemic sclerosis.
Evolution of the molecular profiles (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing]) of systemic sclerosis during 5 years. | 5 years
  This study is descriptive (non-analytical), without prior hypothesis. Molecular profiles will be assessed by integration of multi-OMIC tools from a wide range of areas of biochemistry, chemistry, physics, computing science and molecular biology.
  During the 5-year follow-up, the investigating physician will remain attentive to the appearance of a new clinical element which will mark the course of the systemic sclerosis.
Evolution of the molecular profiles (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing]) of inflammatory myopathies during 5 years. | At Day 1
  This study is descriptive (non-analytical), without prior hypothesis. Molecular profiles will be assessed by integration of multi-OMIC tools from a wide range of areas of biochemistry, chemistry, physics, computing science and molecular biology.
  During the 5-year follow-up, the investigating physician will remain attentive to the appearance of a new clinical element which will mark the course of the inflammatory myopathies.
Evolution of the molecular profiles (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing]) of inflammatory myopathies during 5 years. | At 12 months
  This study is descriptive (non-analytical), without prior hypothesis. Molecular profiles will be assessed by integration of multi-OMIC tools from a wide range of areas of biochemistry, chemistry, physics, computing science and molecular biology.
  During the 5-year follow-up, the investigating physician will remain attentive to the appearance of a new clinical element which will mark the course of the inflammatory myopathies.
Evolution of the molecular profiles (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing]) of inflammatory myopathies during 5 years. | 5 years
  This study is descriptive (non-analytical), without prior hypothesis. Molecular profiles will be assessed by integration of multi-OMIC tools from a wide range of areas of biochemistry, chemistry, physics, computing science and molecular biology.
  During the 5-year follow-up, the investigating physician will remain attentive to the appearance of a new clinical element which will mark the course of the inflammatory myopathies.
Comparison of the molecular profiles between systemic sclerosis and inflammatory myopathies at disease early stage. | Day 1
  Comparison of the molecular profiles (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing] between systemic sclerosis and inflammatory myopathies at disease early stage.
Comparison of the molecular profiles between systemic sclerosis and inflammatory myopathies at one year and versus disease early stage. | At 12 months
  Comparison of the molecular profiles (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing] between systemic sclerosis and inflammatory myopathies at one year and versus disease early stage.
Comparison of the molecular profiles between systemic sclerosis and inflammatory myopathies at 5 years and versus disease early stage. | At 5 years
  Comparison of the molecular profiles (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing] between systemic sclerosis and inflammatory myopathies at 5 years and versus disease early stage.

SECONDARY OUTCOMES:
Identification of molecular profiles specific to the evolution of clinical and biological characteristics of systemic sclerosis and inflammatory myopathies | 5 years
  Study of the molecular profile (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing]) of systemic sclerosis during a systemic or infectious complication (initial profile compared to the profile at the time of the complication)
Identification of molecular profiles specific to the impact of the implementation of targeted treatments in systemic sclerosis and inflammatory myopathies | 5 years
  Study of the molecular profile (i.e., genomic [New Generation Sequencing], transcriptomic [RNA chip], proteomic [mass spectrometry] and identification of cell population [single cell RNA sequencing]) of systemic sclerosis before and after the implementation of targeted treatments (immunomodulators, cell therapies).
Assessment of the presence of discriminating molecular profiles in different tissues (blood, skin, muscle) in systemic sclerosis and inflammatory myopathies | 5 years
  Compare the molecular profiles of blood (serum, PMBC), skin (sclerotic, healthy) and muscle, of early and advanced systemic sclerosis and inflammatory myopathies
Assessment of the presence of discriminating molecular profiles in different cell subpopulations within these tissues (blood, skin, muscle) in systemic sclerosis and inflammatory myopathies | 5 years
  Compare the molecular profiles in different cell subpopulations within blood, skin and muscle tissues by single cell analysis in systemic sclerosis and inflammatory myopathies

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Hautepierre, Strasbourg, Bas-Rhin, France